CLINICAL TRIAL: NCT05805696
Title: Treatment and Mapping of Self-compassion, Perfectionism, Stress, Anxiety and Impostor Phenomenon in Patients With Different Dermatological Diseases and Pain
Brief Title: Treatment and Mapping of Impostor Phenomenon
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Elisabet Nylander, Professor/senior consultant, Umeå University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-01511-01
Record Dates: First submitted 2023-03-09; First posted 2023-04-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Dermatoses; Vestibulodynia; Hyperhidrosis; Pain Syndrome
MeSH Terms: conditions — Skin Diseases; Vulvodynia; Hyperhidrosis; Somatoform Disorders

STUDY DESIGN:
Intervention Model Description: All patients will get the same questionnaires and the same intervention
Masking Description: The participants will get a code to use for all questionnaires. The questionnaires and the intervention messages will be handled by a person that will not be involved in the answers. The questionnaires will be answered on-line with a code and handled by a person not former involved and thus completely unaware of which patients are attending.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment for five weeks (Experimental): The patients will get questionnaires before and 12 weeks and 24 weeks after intervention. The intervention will last for 5 weeks.
  Interventions: Behavioral: Impostor tasks

INTERVENTIONS:
Behavioral: Impostor tasks — Tasks to do every week

SUMMARY:
The aim of this study is to evaluate persons/patients with different skin diseases or pain to evaluate whether unhealthy perfectionism, stress, anxiety, impostor phenomenon (inability to realistically assess your competence and skills) and lack of self-compassion (a positive attitude towards ourselves), have impact on symptoms, handling, and treatment regarding some dermatological diseases/pain.

DETAILED DESCRIPTION:
The investigators have noticed that these conditions are common among patients attending the clinic. The investigators therefore want to do mapping of the occurrence and make an intervention to be able to change and evaluate handling of these patients. The hypothesis is that there is a connection between these conditions and that they are all part of the patients´ disease. The study will be done by using validated questionnaires which are answered anonymously using a code, that is known only by the participant, and with exercises/interventions for five or ten weeks. The questionnaires and interventions are formerly used in several international studies and by the investigators in populations of healthy persons with different professions.

Examples of diseases is localised provoked vulvodynia (former vulvar vestibulitis) a state of pain that mainly affects young women. The symptoms are localized to the vulvar vestibulum and provoked by touch and experienced by the patient as pain or burning. The aetiology is not clearly known but probably due to both physical and psychological factors. Treatment is due to several strategies like treating the pain, rehabilitation of the perineum, and psychosocial support. Persons with this type of pain will also answer a short questionnaire regarding their symptoms. Another example is hyperhidrosis is excessive sweating without known cause. Hyperhidrosis may be primary focal or multifocal with debut in childhood. Secondary hyperhidrosis is often due to another disease. Hyperhidrosis often means big stress on mental health but may also affect physical functions. Persons with hyperhidrosis estimate their quality of life equal with those affected by severe acne or psoriasis.

The investigators´ ongoing research with mapping of these different traits of character shows that the occurrence is increasing, but no treatment has so far been available in Sweden. The investigators therefore want to evaluate whether treatment by intervention with one or two exercises each week may diminish the occurrence of impostor phenomenon and to be able to influence the disease.

The questionnaires that will be used are "Self-Compassion scale short version" (SCS-SF), "Clance Impostor Phenomenon scale" (CIPS), "Perceived Stress scale 4" (PSS-4), "Generalized Anxiety Disorder-2" (GAD-2), and "Clinical Perfectionism Questionnaire short form" (CPQ-SF). These questionnaires are validated by other investigators and used in several international research studies. The questionnaires have already been translated from English to Swedish, except CIPS that has been translated and back-translated. There will also be questions on gender, age, and term. The software for statistical analyses is Statistical Package for the Social Sciences (SPSS) version 27 from International Business Machines Corporation (IBM).

Before starting treatment, the participants will get a web-based survey including twenty questions about impostor phenomenon (CIPS), six questions about stress and anxiety (PSS-4 and GAD-2), twelve questions about self-compassion (SCS-SF) and six questions about perfectionism (CPQ-SF). The questionnaires are repeated week twelve and 24 after intervention. After inclusion and answering the first questionnaire the persons are asked to participate in a series of one or two interventions, 30 minutes each, every week for ten or five weeks respectively.

ELIGIBILITY:
Inclusion criteria

* Patients attending the Dept of Dermatology and Venereology
* Diagnosed with a dermatological disease

Exclusion criteria

* Age under 18
* Not able to read/speak Swedish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-05-15 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Signs of impostor | At the beginning, after 12 and 24 weeks
  Questionnaire regarding impostor
Signs of disease/pain | At the beginning, after 12 and 24 weeks
  Questionnaire regarding symptoms

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Umea University, Umeå
  - Dept of Public Health and Clinical Medicine, Umeå University, Umeå

IPD SHARING:
Plan to Share IPD: No